CLINICAL TRIAL: NCT04656223
Title: Digital Adherence Monitoring of Inhalative Therapy in Real- Life Conditions
Acronym: ADITION
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CQVM149BDE01
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Asthma
Keywords: mobile Health; mHealth; Propeller Health; MF/IND/GLY Breezhaler®; FDC; Fixed dose combination; Mometasone Fuorat; Indacaterol; Glycopyrronium
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- MF/IND/GLY Breezhaler® plus Propeller Health: patients receiving MF/IND/GLY Breezhaler® plus electronic inhalation tracking sensor (Propeller Health) according to label
  Interventions: Combination Product: MF/IND/GLY plus sensor system
- Other FDC therapy: patients receiving ICS+LABA+LAMA FDC therapy according to label
  Interventions: Drug: FDC therapy

INTERVENTIONS:
Combination Product: MF/IND/GLY plus sensor system — There is no treatment allocation. Patients administered MF/IND/GLY plus sensor system by prescription that have started before inclusion of the patient into the study will be enrolled.
  Subjects will receive MF/IND/GLY together with the Propeller add-on sensor for the Breezhaler® according to label.
  Groups: MF/IND/GLY Breezhaler® plus Propeller Health
Drug: FDC therapy — There is no treatment allocation. Patients administered FDC therapy by prescription that have started before inclusion of the patient into the study will be enrolled.
  Groups: Other FDC therapy

SUMMARY:
This study is designed as a multicenter, observational, non-interventional, open label, 26-week study in order to observe how asthma control changes under treatment with Mometasone Fuorat/Indacaterol/ Glycopyrronium (MF/IND/GLY) Breezhaler® sensor system or under treatment with fixed-dose combination (FDC) triple therapy after 26 weeks of treatment.

DETAILED DESCRIPTION:
Subjects in one group will receive MF/IND/GLY together with the Propeller add-on sensor for the Breezhaler® and access to the smartphone app according to label. Subjects in the other group will receive any triple FDC according to label. The physician's decision to initiate or switch a patient to MF/IND/GLY Breezhaler® system or any other triple FDC must have been taken prior to and independently from the decision to include the patient in the study.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, all of the following inclusion criteria must be met:

1. Patients (m/f/d) at the age of ≥18
2. Written declaration of consent
3. Asthma diagnosis according to German Asthma Guideline NVL, 4th edition
4. Suitability for a therapy with MF/IND/GLY in combination with the sensor system or another ICS+LABA+LAMA FDC according to SPC
5. At least 6 months of inhaled therapy with ICS+LABA (high dose) or ICS+LABA+LAMA (medium or high dose) before switching or escalating asthma medication at baseline
6. Change or escalation of the asthma medication to MF/IND/GLY in combination with the sensor system or another ICS+LABA+LAMA FDC according to the therapy decision of the treating physician
7. Availability of at least one ACT value of the last 6 months before consent
8. Cohort treated with MF/IND/GLY in combination with the sensor system

   * Owning an Android or iOS smartphone or tablet on which the app can be installed (via WiFi or mobile data network) and run (requires about 75 megabytes of storage space) and which is capable of establishing a Bluetooth connection to the sensor The patient must agree to activate the app, the Bluetooth connection and the mobile data connection regularly (at least once a month).
   * Availability of an e-mail address

Exclusion Criteria:

To participate in the study, none of the following exclusion criteria must apply:

1. Use of a digital inhaler-coupled inhalation tracking system to support adherence in the last 3 months prior to study entry
2. Simultaneous participation in an interventional study or in another Novartis-sponsored noninterventional study
3. Asthma therapy with a biological agent, if not stable at the same dosage for at least 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from approximately 25 pulmonology centers across Germany.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change in asthma control test (ACT) score | Baseline, week 26
  ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control.
  It is a self-administered questionnaire comprising five items that are assessed on a five point categorical scale (1 to 5) and the scores are summed to give a total score ranging from 5 to 25, with a score of >=20 denoting 'controlled asthma', a score of 16-19 denoting 'partially controlled asthma', and a score of <=15 denoting 'uncontrolled asthma'. The total score is calculated as the sum of the scores from all 5 questions. Higher scores indicates improved asthma control.

SECONDARY OUTCOMES:
Description of reasons for prescribing MF/IND/GLY plus sensor or triple FDC as indicated by the physician | Baseline
  Description of reasons for prescribing MF/IND/GLY plus sensor or triple FDC as indicated by the physician will be provided
Description of of patient characteristics at baseline | Baseline
  Description of patient characteristics at baseline in the treatment groups receiving MF/IND/GLY plus sensor or triple FDC will be provided
Percentage of patients showing an improvement in self-reported test adherence to inhalers (TAI) questionnaire | 26 weeks
  TAI test is a 12-item questionnaire designed to assess the adherence to inhalers in patients with asthma.
  Ten questions are answered by the patients, and have to rate each question from 1 to 5. Total score can go between 10 and 50; 50 points correlates to "adherent", 46-49 points correlates to "moderate adherent" and lower than 45 points correlate to "not adherent".
  Two additional questions are answered by the physician
Course of adherence in the subgroup receiving MF/IND/GLY plus sensor | 26 weeks
  Adherence course according to inhalation tracking data in the subgroup treated with MF/IND/GLY plus sensor will be provided
Percentage of days with adherence to treatment in the subgroup receiving MF/IND/GLY plus sensor | 26 weeks
  Percentage of days with adherence to treatment in the subgroup receiving MF/IND/GLY plus sensor will be provided
Percentage of patients achieving the minimal clinically important difference (MCID) change | Baseline, week 26
  Percentage of patients achieving the minimal clinically important difference (MCID) change from baseline ACT ≥ 3 points will be provided
Percentage of patients with an ACT score <19 | 26 weeks
  Percentage of patients with an ACT score of <19 at baseline and following 26 weeks will be provided
Change in Post-dose trough Forced Expiratory Volume in one second (FEV1) | Baseline, week 26
  FEV 1 it is the amount that is exhaled in the first second of purposefully trying to breathe out as much air as possible.
Change in Forced vital capacity (FVC) | Baseline, week 26
  FVC is the volume of air that can forcibly be blown out after full inspiration, measured in liters.
Adverse events | 26 weeks
  Adverse events will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Germany (22):
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Braunschweig, Lower Saxonia
  - Novartis Investigative Site, Hanover, Lower Saxonia
  - Novartis Investigative Site, Ibbenbueren, Rhineland-Palatinate
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Ansbach
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Sachsa
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Burgwedel
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Fürstenwalde
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Radebeul
  - Novartis Investigative Site, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CQVM149BDE01 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18137